CLINICAL TRIAL: NCT04131296
Title: Association of Lung Bacteriobiota With Intensive Care Unit Mortality in ARDS Patients: MicroFlu Study
Brief Title: Lung Bacteriobiota and Influenza Mortality
Acronym: MicroFlu
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Dr Pauline Esteves, Doctor, University of Bordeaux
Other Study IDs: MicroFlu
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Influenza; Critical Illness
Keywords: influenza; microbiota; intensive care unit
MeSH Terms: conditions — Influenza, Human; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum or tracheal aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: influenza screening — positive influenza screening

SUMMARY:
Influenza is a potentially lethal disease still responsible for thousands excess deaths both in Europe and the United States. Despite the use of neuraminidase inhibitors, its treatment is mostly based on symptomatic care. Lung microbiota has been shown to be involved in the immunity against influenza and is correlated with lung inflammation in numerous chronic respiratory diseases. We therefore aim to analyse the correlation between lung bacteriobiota and influenza ICU mortality

DETAILED DESCRIPTION:
Influenza is a viral disease which is still responsible for thousands of excess deaths par year both in Europe and in the US. Despite the use of neuraminidase inhibitors, its treatment is mostly based on symptomatic care. As lung microbiota is correlated with lung inflammation in numerous chronic respiratory diseases, we hypothesize that lung microbiota would be correlated with influenza outcomes. In a pilot study, we found that lung bacteriobiota but not mycobiota is associated with influenza ICU mortality. We therefore aim to confirm this correlation between lung bacteriobiota and influenza mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 year-old admitted to intensive care unit
* Influenza diagnosis by PCR or rapid diagnostic test

Exclusion Criteria:

* Guardianship or curatorship
* Prisoners
* No health insurance
* No legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Influenza patients admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Lung bacteriobiota and ICU mortality | at admission
  Comparison of lung bacteriobiota alpha diversity between influenza ICU survivors and non-survivors

SECONDARY OUTCOMES:
Lung bacteriobiota and ICU mortality | at admission
  Analysis of lung bacteriobiota beta diversity between influenza ICU survivors and non-survivors
Lung bacteriobiota and 7-day mortality | at admission
  Analysis of lung bacteriobiota beta diversity between influenza 7-day survivors and non-survivors
Bacteria and ICU mortality | at admission
  Association of bacteria with influenza ICU mortality by LefSe method
Bacteria and 7-day mortality | at admission
  Association of bacteria with influenza 7-day mortality by LefSe method
ICU mortality based on Shannon index | at admission
  Comparison of ICU mortality based on a threshold of 1.79 for Shannon Index
Lung bacteriobiota and 7-day mortality | at admission
  Comparison of lung bacteriobiota alpha diversity between influenza 7-day survivors and non-survivors

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Medical intensive care unit, Pellegrin hospital, Bordeaux, Nouvelle-Aquitaine
  - Intensive care unit, CH Robert Boulin, Libourne
  - Intensive care unit, CH Francois Mitterrand, Pau

IPD SHARING:
Plan to Share IPD: No